CLINICAL TRIAL: NCT04776850
Title: Pre-Transplant Immunosuppression and Related Haploidentical Hematopoietic Cell Transplantation for Patients With Severe Hemoglobinopathies
Brief Title: Pre-transplant Immunosuppression and Donor Stem Cell Transplant for the Treatment of Severe Hemoglobinopathies
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Competing protocol opened in Adult SCT that will include pediatric patients and is now multi-center. No patients enrolled on study.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0952; NCI-2021-00365 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0952 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-03-02 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2022-11

CONDITIONS: Beta Thalassemia Major; Sickle Beta 0 Thalassemia; Sickle Beta Plus Thalassemia; Sickle Beta Thalassemia; Sickle Cell Disease; Sickle Cell-SS Disease
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell | interventions — Bortezomib; Busulfan; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Plasmapheresis; Plasma Exchange; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PTIS, HCT) (Experimental): See Detailed Description.
  Interventions: Drug: Bortezomib; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Biological: Lapine T-Lymphocyte Immune Globulin; Drug: Mycophenolate Mofetil; Procedure: Plasmapheresis; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-Thymocyte Globulin Rabbit; Grafalon; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; rATG; Thymoglobulin
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: CellCept; MMF
Procedure: Plasmapheresis — Undergo plasmapheresis
  Other Names: Plasma Exchange; Therapeutic Plasma Exchange; Therapeutic Plasmapheresis
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This clinical trial studies the effect of pre-transplant immunosuppression (PTIS) and donor stem cell transplant in treating patients with severe blood diseases (hemoglobinopathies). PTIS helps prepare the body for the transplant and lowers the risk of developing graft versus host disease (GVHD). Hematopoietic cells are found in the bone marrow and produce blood cells. Hematopoietic cell transplantation (HCT) injects healthy hematopoietic cells into the body to support blood cell production. PTIS and HCT may help to control severe hemoglobinopathies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate event-free survival (EFS) at 2-years post HCT.

SECONDARY OBJECTIVES:

I. Assess event-free survival (EFS) at 100 days and 1 year post HCT. II. Assess overall survival (OS) at 100 days and 1 year post HCT. III. 30-day transplant-related mortality (TRM). IV. Time to platelet and neutrophil engraftment. V. Rate of graft failure (primary and secondary) through day 100. VI. Incidence of acute graft-versus-host disease (aGVHD) by day 100. VII. Incidence of chronic graft-versus-host disease (cGVHD) by 1 year and 2 years.

VIII. Rate of grade II or greater organ toxicity through day 100. IX. Incidence of hepatic sinusoidal obstruction syndrome (SOS) by day 100. X. Incidence of central nervous system (CNS) toxicities including posterior reversible encephalopathy syndrome (PRES) by day 100.

XI. Incidence of infectious complications through day 100.

EXPLORATORY OBJECTIVES:

I. Effect of HCT on clinical and laboratory manifestations of hemoglobinopathies by 1 and 2 years after HCT.

II. Assess the pharmacokinetic profile of busulfan and thymoglobulin to better understand post-transplant outcomes.

III. Assess immune reconstitution kinetics post HCT.

OUTLINE:

DONOR-SPECIFIC ANTI-HLA DESENSITIZATION: Patients with donor-specific anti-HLA antibody titers >= 1:3,000 at the start of PTIS receive rituximab intravenously (IV) on days -69, -41, -28, and -13 and bortezomib IV over less than 1 minute on days -68, -65, -40, and -37 in the absence of unacceptable toxicity. Patients with donor-specific anti-HLA antibody titers > 1:15,000 at the start of PTIS receive receive rituximab IV on days -69, -41, -28, and -13 and bortezomib IV over less than 1 minute on days -68, -65, -62, -58, -40, -37, -34, and -31 in the absence of unacceptable toxicity. Patients with donor-specific anti-HLA antibody titers > 1:5,000 at the start of conditioning may also undergo plasmapheresis on day -12.

PTIS: Patients receive fludarabine phosphate (fludarabine) IV over 1 hour and dexamethasone IV over less than 1 minute on days -68 to -64 and days -40 to -36 in the absence of disease progression or unacceptable toxicity.

CONDITIONING: Patients receive lapine T-lymphocyte immune globulin (rATG) IV over 4-6 hours on days -12 to -10, fludarabine phosphate IV over 1 hour on days -8 to -4, and busulfan IV over 2 hours on days -7 to -4 in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: Patients undergo HCT on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 2-3 hours on days 3 and 4 in the absence of unacceptable toxicity. Beginning on day 5, patients also receive tacrolimus IV continuously daily and then orally (PO) twice daily (BID) at the discretion of the treating physician for up to 12 months, and mycophenolate mofetil IV or PO BID up to day 60 in the absence of unacceptable toxicity.

After completion of HCT, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2-30 years-of-age with confirmed sickle cell disease (SCD) (SS & sickle beta [SB]-thalassemia, both sickle beta 0 [SB0] and sickle beta plus [SB+]) or severe B-thalassemia major are potentially eligible
* Patients with SCD should also meet the following eligibility criteria as outlined by the Center for Medicaid and Medicare Services: sickle cell disease and at least one of the following:

  * Stroke or neurological deficit lasting > 24 hours
  * Recurrent acute chest syndrome (ACS): 2 or more episodes of ACS in 2-year period preceding enrollment
  * Recurrent vaso-occlusive pain crises: 3 or more episodes per year in 2-year period preceding enrollment or recurrent priapism (3 or more episodes in the 2 years preceding enrollment)
  * Chronic transfusion program defined as 8 or more packed red blood cells (PRBC) transfusions per year to prevent central nervous system and/or vaso-occlusive complications in 1-year period preceding enrollment
  * Impaired neuropsychological function and abnormal cerebral magnetic resonance imaging (MRI) scan (silent strokes)
  * Stage I or II sickle lung disease
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate 30-50% of predicted normal value)
  * Bilateral proliferative retinopathy and major visual impairment in at least one eye
  * Osteonecrosis of multiple joints
  * Echocardiographic finding of tricuspid valve regurgitant jet velocity (TRJV) >= 2.7 m/sec
* Patients with B-thalassemia are considered as severe if they are/have any of the following:

  * Transfusion-dependent
  * Evidence of extra-medullary hematopoiesis
  * Pesaro Class III
* Patients shall not proceed to HCT without confirmation of primary diagnosis by review of available newborn screening results or hemoglobin electrophoresis and/or genetic testing
* DONOR: High resolution HLA typing will be performed on all willing and available biologic parents and siblings without clinically significant hemoglobinopathy. Preference will be given to donors with the lowest number of HLA-allele mismatches
* DONOR: Donor-specific anti-HLA antibodies will be obtained and analyzed from all patients. Preference will be given to donors with absent or low titer anti HLA-donor specific antibody levels when possible

Exclusion Criteria:

* Uncontrolled infection
* Females who are pregnant and/or unwilling to cease breastfeeding
* Seropositivity for human immunodeficiency virus (HIV)
* Lansky or Karnofsky performance status < 70%
* Life expectancy severely limited by concomitant illness
* Uncontrolled arrhythmias or symptomatic cardiac disease
* Uncontrolled symptomatic pulmonary disease
* Evidence of chronic active hepatitis or cirrhosis
* Serum conjugated (direct) bilirubin > 2 x upper limit of normal for age. Participants are not excluded if the serum conjugated (direct) bilirubin is > 2 x the upper limit of normal for age as per local laboratory and:

  * There is evidence of a hyperhemolytic reaction after a recent red blood cell (RBC) transfusion, OR
  * There is evidence of moderate direct hyperbilirubinemia defined as direct serum bilirubin < 5 times upper limit of normal (ULN) and not caused by underlying hepatic disease
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 5 x upper limit of normal for age
* Serum creatinine > 1.5 x upper limit of normal for age AND estimated or measure creatinine clearance < 70 mL/min/1.72 m^2
* Patient, parent or guardian unable/unwilling to provide consent and when indicated, assent
* Patients with available HLA-matched related donor
* Prior receipt of gene therapy
* DONOR: All potential donors shall be tested by hemoglobin electrophoresis. Any potential donor with a clinically significant hemoglobinopathy will be deemed ineligible. Donors with sickle cell trait and beta thalassemia trait are eligible to donate

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | At 2 years post-hematopoietic cell transplantation (HCT)
  EFS is defined as survival time following HCT without a qualifying event. Will be summarized by the Kaplan-Meier method with 95% confidence intervals.

SECONDARY OUTCOMES:
Event-free survival | Up to 100 days post-HCT
  EFS is defined as survival time following HCT without a qualifying event. Will be summarized by the Kaplan-Meier method with 95% confidence intervals.
Event-free survival | Up to 1 year post-HCT
  EFS is defined as survival time following HCT without a qualifying event. Will be summarized by the Kaplan-Meier method with 95% confidence intervals.
Overall survival | Up to 100 days post-HCT
  Will be summarized by the Kaplan-Meier method.
Overall survival | Up to 1 year post-HCT
  Will be summarized by the Kaplan-Meier method.
Transplant-related mortality | Up to 30 days post-HCT
  Will be summarized by the Kaplan-Meier method.
Time to platelet and neutrophil engraftment | Up to 2 years post-HCT
  Will be estimated using the method of Gooley et al.
Incidence of graft failure (primary and secondary) | Up to 100 days post-HCT
  Will be estimated using the method of Gooley et al.
Incidence of acute graft-versus-host disease | Up to 100 days post-HCT
  Will be estimated using the method of Gooley et al.
Incidence of chronic graft-versus-host disease | Up to 1 year post-HCT
  Will be estimated using the method of Gooley et al.
Incidence of chronic graft-versus-host disease | Up to 2 years post-HCT
  Will be estimated using the method of Gooley et al.
Incidence of grade II or greater organ toxicity | Up to 100 days post-HCT
  Will be reported as counts with percentages.
Incidence of hepatic sinusoidal obstruction syndrome | Up to 100 days post-HCT
  Will be reported as counts with percentages.
Incidence of central nervous system toxicities including posterior reversible encephalopathy syndrome | Up to 100 days post-HCT
  Will be reported as counts with percentages.
Incidence of infectious complications | Up to 100 days post-HCT
  Will be reported as counts with percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Kris M Mahadeo, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT04776850/ICF_000.pdf